CLINICAL TRIAL: NCT03186495
Title: Investigation of Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Multiple Doses of Somapacitan in Subjects With Various Degrees of Impaired Renal Function Compared to Subjects With Normal Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN8640-4297; U1111-1187-9141 (Other: World Health organization (WHO)); 2016-003910-29 (Registry Identifier: EudraCT)
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Growth Hormone Disorder; Adult Growth Hormone Deficiency; Growth Hormone Deficiency in Children
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — somapacitan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Normal renal function (Experimental): Subjects with normal renal function
  Interventions: Drug: Somapacitan
- Mild renal impairment (Experimental): Subjects with mild renal impairment
  Interventions: Drug: Somapacitan
- Moderate renal impairment (Experimental): Subjects with moderate renal impairment
  Interventions: Drug: Somapacitan
- Severe renal impairment (Experimental): Subjects with severe renal impairment
  Interventions: Drug: Somapacitan
- Requiring haemodialysis treatment (Experimental): Subjects requiring haemodialysis treatment
  Interventions: Drug: Somapacitan

INTERVENTIONS:
Drug: Somapacitan — All subjects will receive three (0.08 mg/kg) consecutive once-weekly s.c. (under the skin) administrations of somapacitan

SUMMARY:
The trial is conducted in Europe. The aim of the trial is to investigate the steady state exposure of somapacitan in subjects with various degrees of renal impairment (mild, moderate, severe renal impairment, requiring haemodialysis treatment) compared to subjects with normal renal function

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-75 years (both inclusive) at the time of signing informed consent
* Body mass index between 18.5-34.9 kg/sqm (both inclusive)
* Meeting the pre-defined glomerular filtration rate for any of the renal function groups 1-4 (based on the measured glomerular filtration rate using exogenous sinistrin (Inutest®) as a filtration marker) or being in treatment with haemodialysis

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method (adequate contraceptive measure as required by local regulation or practice). Male of reproductive age who or whose partner(s) is not using adequate contraceptive methods (adequate contraceptive measures as required by local regulation or practice) or male who is not willing to refrain from donating semen for at least 16 days after last trial product administration
* Any disorder, except for conditions associated with renal impairment in the groups of subjects with reduced renal function, which in the investigator's opinion might jeopardise subject's safety, evaluation of results, or compliance with the protocol. For example, arterial hypertension, anaemia, impaired glucose tolerance or type 2 diabetes are accepted in the group of subjects with renal impairment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2018-05-17 (Actual); Study Completion 2018-05-17 (Actual)

PRIMARY OUTCOMES:
Area under the somapacitan serum concentration time curve | From time 0 to 168 hours after the last dosing on Day 15.
  Calculated based on the serum concentrations measured in ug/l

SECONDARY OUTCOMES:
Maximum serum concentration of somapacitan | After the last dosing on Day 15 up until Day 43
  Measured in ng/ml
Time to maximum serum concentration of somapacitan | After the last dosing on Day 15 up until Day 43
  Calculated based on the serum concentrations measured in ug/l
Incidence of adverse events | Day 0 - 43
  Count and % of events
Occurrence of anti-somapacitan antibodies | Day 0 - 43
  Count or % of events

CONTACTS AND LOCATIONS:
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Derived] Bentz Damholt B, Dombernowsky SL, Dahl Bendtsen M, Bisgaard C, Hojby Rasmussen M. Effect of Kidney or Hepatic Impairment on the Pharmacokinetics and Pharmacodynamics of Somapacitan: Two Open-Label, Parallel-Group Trials. Clin Pharmacokinet. 2021 Aug;60(8):1015-1027. doi: 10.1007/s40262-021-00990-7. Epub 2021 Mar 23. PMID 33754315